CLINICAL TRIAL: NCT05419180
Title: Study of the Interest of the Combination of Stiripentol (Diacomit®) and Carbamazepine in the Treatment of Patients With Pharmacoresistant Focal Epilepsies
Brief Title: Study of Interest of Stiripentol and Carbamazepine in the Treatment of Patients With Pharmacoresistant Focal Epilepsies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARBASTIR (STP225)
Record Dates: First submitted 2022-05-16; First posted 2022-06-15 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2022-05

CONDITIONS: Pharmacoresistant Focal Epilepsies
MeSH Terms: interventions — stiripentol

STUDY DESIGN:
Intervention Model Description: retrospective part and prospective part
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stiripentol (Other)
  Interventions: Drug: Stiripentol

INTERVENTIONS:
Drug: Stiripentol — Since the treatment usually received by patients should not be modified, the sponsor will not intervene in any way in the therapeutic management of patients.

SUMMARY:
This is a monocentric, open-label clinical study, presenting a retrospective part and a prospective part, studying the data of patients with drug-resistant focal epilepsies and treated with the combination of stiripentol (Diacomit®) and Carbamazepine.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective part of the research:

The medical records of CRéER patients with the following criteria will be included in the retrospective part of the research by an investigator:

1. With pharmacoresistant epilepsy, i.e. a history of failure of two well-conducted and well-tolerated antiepileptic treatment regimens, either as monotherapy or as combination therapy,
2. Receiving or having received a treatment combining stiripentol and carbamazepine for a period of at least 15 days,
3. Having at least one evaluation data after the initiation of treatment with stiripentol and carbamazepine (a follow-up visit after the initiation of the study treatment),
4. For which an information note indicating the possibility of opposing the processing of data has been provided.

   * Prospective part of the research:

Among the patients whose medical records are included in the retrospective part of the research, those who meet the following criteria will be able to participate in the prospective part of the research:

1. Currently treated with stiripentol in combination with carbamazepine for at least 15 days and still being followed in the center,
2. Weighing at least 5 kg (minimum weight in accordance with the blood volume taken),
3. Having read, or whose parents have read, the information note and signed the consent form. For children, if their level of understanding allows it, their consent will also be sought,
4. Having sufficient knowledge, or whose parents or legal guardians have sufficient knowledge, of the French language to read, understand and complete the research documents,
5. Members or beneficiaries of a social security scheme. These patients, both children and adults, will be welcomed at the CIC.

Exclusion Criteria:

- Retrospective part of the research : Patients objecting to the collection of their data will not participate in the research.

- Prospective part of the research :

Patients with the following criteria will not be able to participate in the prospective part of the research:

1. Participating simultaneously in another interventional clinical trial or in a period of exclusion following a previous trial,
2. Whose state of health does not allow him to give his consent,
3. Under guardianship or curatorship,
4. Under judicial protection or person deprived of liberty.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Age | through study completion, an average of 1 year
  Age of onset, nature of the first seizure and description of the type of the first seizure.
Previous antiepileptic treatments received | through study completion, an average of 1 year
  proportion of patients having received each antiepileptic treatment; for the treatments received, description of the reasons for stopping.
Surgery | through study completion, an average of 1 year
  proportion of patients having undergone epilepsy surgery.
Adjustment of carbamazepine treatment over the time | through study completion, an average of 1 year
  mean and median duration of treatment, mean and median daily dose received, dose change(s) during treatment...
Adjustment of stiripentol treatment over the time | through study completion, an average of 1 year
  mean and median duration of treatment, mean and median daily dose received, dose change(s) during treatment...
Adjustment of concomitant treatments over the time | through study completion, an average of 1 year
  continuation without change, change in dosage, discontinuation
monthly seizures over the time | through study completion, an average of 1 year
  description of the average number of monthly seizures since the last visit (total and by type of seizure)
status epilepticus in the past | through study completion, an average of 1 year
  proportion of patients who presented with status epilepticus
duration of the status epileticus over the time | through study completion, an average of 1 year
  duration of status epilepticus
emergency room consultation and/or hospitalization over the time | through study completion, an average of 1 year
  Proportion of patients requiring an emergency room consultation and/or hospitalized during the period preceding the visit.
emergency antiepileptic treatment over the time | through study completion, an average of 1 year
  Proportion of patients taking emergency antiepileptic treatment in the period before each visit
frequency of the status epileticus over the time | through study completion, an average of 1 year
  frequency of status epilepticus

SECONDARY OUTCOMES:
Retention rate of the combination | through study completion, an average of 1 year
  The retention rate of the combination will correspond to the proportion of patients still receiving the combination (carbamazepine and stiripentol) at a given time.
Response to the combination | through study completion, an average of 1 year
  The rate of patients responding to the combination will be defined by the percentage of patients in whom a 50% reduction in visible seizures will be observed since the initiation of the carbamazepine and stiripentol combination.
  Will be estimated:
  oThe percentage of responder patients at the post-initiation visit of the combination (first follow-up visit after initiation of stiripentol) oThe percentage of responder patients during treatment regardless of the duration of treatment after which the response is obtained.
  oThe cumulative incidence of responder patients.
Tolerance of the combination. | through study completion, an average of 1 year
  Proportion of patients with Adverse Effects (AEs) related to the combination or to one of the treatments,
Frequency and nature of the adverse events over the time | through study completion, an average of 1 year
  Frequency and nature of the adverse events over the time
Abnormal biological parameters (NFS and liver) | through study completion, an average of 1 year
  proportion of patients with abnormal laboratory values (NFS and liver function) during

OTHER OUTCOMES:
Maximum Concentration (Cmax) for stiripentol, carbamazepines and its metabolites | through study completion, an average of 1 year
  Cmax calculation
Area under the plasma concentration versus time curve (AUC) 0-8 for stiripentol, carbamazepines and its metabolites | through study completion, an average of 1 year
  AUC0-8 calculation
Area under the plasma concentration versus time curve (AUC) 0-24 for stiripentol, carbamazepines and its metabolites | through study completion, an average of 1 year
  AUC0-24 calculation
Time of Maximum (Tmax)concentration for stiripentol, carbamazepines and its metabolites | through study completion, an average of 1 year
  Tmax calculation
half-life (t1/2) for stiripentol, carbamazepines and its metabolites | through study completion, an average of 1 year
  t1/2 calculation
Pre-dose trough concentration (Ctrough) for stiripentol, carbamazepines and its metabolites | through study completion, an average of 1 year
  Ctrough calculation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence Epilepsies Rares / Centre Investigation Clinique (CIC) - Hôpital Necker-Enfants Malades, Paris, France